CLINICAL TRIAL: NCT04755855
Title: Sinonasal Cancer Study to Evaluate Oncologic Outcomes and Quality of Life
Brief Title: Prospective Sinonasal Cancer Multi-institution Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jacob G. Eide, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 20-010181
Record Dates: First submitted 2021-02-09; First posted 2021-02-16 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Sinonasal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a multi-institution prospective study of patients with sinonasal malignancies. The goal of this study is to learn more about the course of sinonasal cancer, treatment outcomes, and patient quality of life. In addition, central mutational and genomic analysis of tumor tissue will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 30 days (non-inclusive) and 99 years (inclusive)
* Patients with a diagnosis of sinonasal cancer
* Patients undergoing treatment at Mayo Clinic

Exclusion Criteria:

* Healthy individuals
* Unwilling to sign the informed consent

Ages: 30 Days to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing treatment for sinonasal cancers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Oncologic outcomes as measured by overall survival, disease specific survival and recurrence free survival | Through study completion, an average of 5 years

SECONDARY OUTCOMES:
Quality of life outcomes including the University of Washington Quality of Life Questionnaire (UW-QOL v4) and the Sinonasal Outcome Test 22 (SNOT22) | Through study completion, an average of 5 years
Describe the molecular foundation of sinonasal malignancies utilizing RNA sequencing to identify transcriptomic tumor profiles | Through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jake Eide, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States